CLINICAL TRIAL: NCT04652921
Title: The Effects of 6-month Supplementation With Creatine and Guanidinoacetic Acid on Biomarkers of Sarcopenia in Elderly
Brief Title: Creatine-Guanidinoacetic Acid Supplementation for Sarcopenia (CREGAAS)
Acronym: CREGAAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DS-04/2020
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine-guanidinoacetic acid (Experimental): 2 grams of creatine and 2 grams of GAA Administered one dose two times per day on an empty stomach in the morning and at the evening
  Interventions: Dietary Supplement: Creatine-guanidinoacetic acid
- Inulin (Placebo Comparator): 4 grams of inulin Administered one dose two times per day on an empty stomach in the morning and at the evening
  Interventions: Other: Inulin

INTERVENTIONS:
Dietary Supplement: Creatine-guanidinoacetic acid — A dietary supplement provided as powder dissolved in a glass of water
  Arms: Creatine-guanidinoacetic acid
Other: Inulin — A dietary supplement provided as powder dissolved in a glass of water
  Arms: Inulin

SUMMARY:
Sarcopenia-driven brain and muscle creatine deficit could be seen as a distinctive pathological facet of this condition, and this might be approached with targeted therapies in aim to restore creatine homeostasis in target tissues. Among potential therapeutic candidates, guanidinoacetate (GAA) appears recently as a direct precursor of creatine that may favorably upregulate muscle and brain creatine concentration. Interestingly, GAA-creatine mixture was found to be superior than creatine itself to effectively improves bioenergetics in the human brain and muscle in healthy humans, perhaps due to the unique transportability features of this combination. Here, we plan to evaluate does creatine-GAA supplementation affects various biomarkers of sarcopenia in elderly.

ELIGIBILITY:
Inclusion Criteria:

* Age > 70 years
* Free of acute disorders

Exclusion Criteria:

* History of dietary supplement use during the past 4 weeks

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in muscular strength | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months

SECONDARY OUTCOMES:
Change in muscle mass | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months
Change in muscle metabolites evaluated with MR spectroscopy | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months
Change in cognitive performance evaluated with Mini-Mental State Exam test | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months
Change in serum creatine | Baseline vs. 6 months post-intervention
  Baseline vs. 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Bioenergetics Lab at Faculty of Sport and PE, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No